CLINICAL TRIAL: NCT05913882
Title: Combined Respiratory Training to Improve Pulmonary and Cough Function in Persons With ALS
Brief Title: Combined Respiratory Training in Persons With ALS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lauren Tabor Gray, PhD, Principal Investigator, Nova Southeastern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL220099
Record Dates: First submitted 2023-05-22; First posted 2023-06-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: ALS; Respiratory Insufficiency; Dysphagia
Keywords: Breathing; Swallowing; Exercise; Bulbar
MeSH Terms: conditions — Respiratory Insufficiency; Deglutition Disorders; Respiratory Aspiration; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lung Volume Recruitment +Expiratory Muscle Strength Training (Experimental): All enrolled participants will commence a combined lung volume recruitment and expiratory muscle strength training exercise regimen following a 5-week no-intervention lead-in period.
  Interventions: Device: Respiratory Muscle Strength Training (LVR+EMST)

INTERVENTIONS:
Device: Respiratory Muscle Strength Training (LVR+EMST) — Combined respiratory muscle strength training regimen that will be completed daily for 5 weeks.

SUMMARY:
The goal of this interventional trial is to learn about lung volume recruitment (LVR) and expiratory muscle strength training (EMST) in a total of up to 39 patients diagnosed with ALS. The following aims will be addressed:

1. Determine the impact of combined LVR and EMST on cough strength and respiratory function in individuals with ALS.
2. Determine the impact of combined LVR and EMST on patient-reported dyspnea and bulbar impairment.
3. Describe the effect of combined LVR and EMST on patient- and caregiver reported burden and quality of life.

DETAILED DESCRIPTION:
In this delayed start, repeated-measures design, pALS will serve as their own control to provide treatment to all participants and control for disease heterogeneity (i.e., interparticipant differences). Participation will include three in-person evaluations and four weekly telehealth therapy sessions (Figure 3). Weekly telehealth therapy sessions will include home peak cough flow assessment, LVR and EMST training sessions to ensure treatment fidelity, maximum phonation time as a surrogate measure of forced vital capacity, and patient-reported outcomes including the ALS Respiratory Symptom Scale. To assess peak cough flow at home, participants will be provided with a commercially available peak cough flow meter (MiniWright, PF100) for guided assessment during telehealth appointments.

Study Timeline.

Study assessments and procedures at each time point are briefly described below and depicted in Table 1.

Screening/Baseline 1 (Week -5).

Following consenting and screening procedures, study personnel will complete the initial baseline assessment procedures. Participants will complete the initial baseline assessment in approximately 60-90 minutes.

Baseline 2 (Week 0).

The Baseline 2 appointment will consist of the identical assessment procedures conducted in the same order as Baseline 1. LVR and EMST training will be introduced and the first training session will be completed during the appointment. Participants will complete the Baseline 2 appointment in ~100-120 minutes.

Telehealth Appointments (Active Training Weeks 0-5).

Weekly telehealth therapy appointments will be conducted during the active training period using the Zoom platform (Zoom Video Communications, Inc). During these sessions, the research clinician will lead a LVR and EMST training session with the participant, complete peak cough flow and maximum sustained phonation testing, and administered surveys including the ALS Functional Rating Scale- Revised and the ALS Respiratory Symptom Scale. Surveys will be screen shared with the participants and data will be recorded on the source documents by the research clinician.

Final Evaluation (Week 5).

The Final Evaluation appointment will consist of the identical assessment procedures conducted in the same order as Baseline 2.

Follow-up Period (6-months).

The follow-up period consists of monthly telehealth visits with the research clinician. Participants who complete the initial 10-week study period will be asked to participate in follow-up. These telehealth visits will include peak cough flow and maximum phonation time assessments, and clinician-administered surveys. During this period, treatment adherence will be tracked using the same daily treatment logs, which will be reviewed during monthly appointments.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of probable or definite ALS in accordance with the Revisited El-Escorial Criteria.
2. Disease duration from symptom onset of ≤ 2 years,
3. Lung volume recruitment and expiratory muscle strength training naïve,
4. Reduced peak cough flow (% predicted for age and gender).

Exclusion Criteria:

1. History of stroke, head and neck cancer or other concomitant disorder that might contribute to dysphagia or respiratory impairment.
2. Use of prescription cough assist or non-invasive volume ventilation devices.
3. Enrollment in another research investigation that might impact cough or respiratory function.
4. Diagnosis of frontotemporal dementia or advanced cognitive impairment.
5. Tracheostomy placement/Use of invasive mechanical ventilation.
6. Contraindications for respiratory training (i.e., history of pneumothorax, severe chronic obstructive pulmonary disease).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Peak Cough Flow | From Baseline 1 to Final Evaluation (10 weeks)
  Greatest cough measurement measured in liters/minute.

SECONDARY OUTCOMES:
Cough Spirometry | From Baseline 2 to Final Evaluation (5 weeks)
  Airflow parameters will be collected during voluntary cough production. The primary outcome obtained from voluntary cough spirometry will be cough volume acceleration (L/s/s), which is an aggregation of peak expiratory flow rate and peak expiratory rise time.
Pulmonary Function Assessment | From Baseline 1 to Final Evaluation (10 weeks)
  Vital capacity with and without LVR. Forced vital capacity will be assessed before and after lung volume recruitment and the measurements will be used to determine the difference between FVC and FVC LIC (% predicted age/gender).
Pulmonary Function Assessment | From Baseline 1 to Final evaluation (10 weeks)
  Maximum respiratory pressure will be obtained to assess inspiratory and expiratory muscle strength (cmH20).
Pulmonary Function Assessment | From Baseline 1 to Final evaluation (10 weeks)
  Maximum phonation time involves the participant sustaining the vowel /ah/ for as long as possible (seconds).

OTHER OUTCOMES:
ALS Functional Rating Scale-Revised (ALSFRS-R, Cedarbaum et al., 2011) | From Baseline 1 to Final Evaluation (10 weeks)
  The ALSFRS-R is the validated, gold standard survey assessing ALS symptom and disease progression to determine disease severity ranging from 0 (severe disease symptomology) to 48 (no overt symptoms)
Center for Neurological Study-Bulbar Function Scale (CNS-BFS, Smith et al., 2011) | From Baseline 1 to Final Evaluation (10 weeks)
  The CNS-BFS is a 21-item validated, patient-reported scale indexing degree of bulbar dysfunction in the domains of speech, salivation and swallowing.

CONTACTS AND LOCATIONS:
Overall Officials: Magalie Thomas, MBA, Study Chair — Nova Southeastern University
Locations (1):
- Nova Southeastern University, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with credentialed individuals upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Following close out of study.
Access Criteria: Please contact the PI Dr Lauren Tabor Gray at Lgray1@nova.edu

REFERENCES:
- See also: Nova ALS Clinic — https://nsuhealth.nova.edu/neuroscience/als.html